CLINICAL TRIAL: NCT05897281
Title: The Effect of SHOOT Exercise Program on Shooting Performance, Muscular Strength and Endurance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Mesken GÜMÜŞSOY, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GU-FTR-MG-01
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2023-07

CONDITIONS: Athletes
Keywords: exercises; muscle strength; shooting; shooters
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: two groups, one control and one exercise group
Who Masked: Outcomes Assessor
Masking Description: the control group will continue their routine training, outcome assesstments will be performed by an investigator who was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): In addition to routine training, the experimental group will be done a progressive resistance band exercise program (SHOOT) created for shooters, 3 days a week for 8 weeks, accompanied by a physiotherapist.
  Interventions: Procedure: SHOOT exercise group
- Control Group (Other): The control group will continue their routine training.
  Interventions: Procedure: routine training group

INTERVENTIONS:
Procedure: SHOOT exercise group — In addition to routine training, the experimental group will be done a progressive resistance band exercise program (SHOOT) created for shooters, 3 days a week for 8 weeks, accompanied by a physiotherapist.
  Arms: Exercise Group
Procedure: routine training group — The control group will continue their routine training
  Arms: Control Group

SUMMARY:
The aim of this study is; to create a special exercise program that will improve the performance of shooting athletes and to examine the effect of this exercise program on shooting performance, muscular strength and endurance of air pistol athletes.

DETAILED DESCRIPTION:
Air pistol shooting is an Olympic sport that requires precise and accurate shooting at the target sign. Many are the factors that can influence performance in Olympic pistol shooting. The ability to stabilize the gun is crucial for performance in Olympic pistol shooting and is thought to be related to the shooters muscular strength. Krasilshchikov, Zuraidee, and Singh suggest that the implementation of a physical conditioning program together with technique training is essential for the improvement of the ability to stabilize the pistol.

Books and journals specialized in Olympic shooting suggest that general physical condition programs, as well as specific strength exercises are necessary in order for performance to be improved. Al Wadi examined the effect of strength exercises on shooting performance and physical parameters with the 8-week station training method with female air pistol shooters in 2015. They found that this exercise program increased arm and waist strength and endurance, the kinetic balance changed positively, and there was a significant correlation between physical variables and shooting performance. However, the study of Belinchon reports that some factors regarding the physical condition of the Spanish Olympic shooters are inferior when compared to athletes of other sports. There is therefore the need for further study on the importance of physical conditioning in Olympic shooting.

ELIGIBILITY:
Inclusion Criteria:

* Athletes who have been shooting air guns for at least 2 years.
* Air pistol athletes between the ages of 17-45.
* Become a licensed shooting athlete.

Exclusion Criteria:

* Any type of musculoskeletal disorder.
* Athletes with a health condition that prevents them from exercising

Ages: 17 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-08-06 (Actual); Study Completion 2023-12-03 (Actual)

PRIMARY OUTCOMES:
Shooting Performance | baseline
  Shooting performance will be calculated with electronic scoring system. (SIUS LS10 Laserscore, Swiss). Electronic Scoring System is an electronic target system for airguns. The target sign at which the shooting is made is 17x17 cm in size; The black dot with a diameter of 11.5 millimeters in the center is 10 points, and the outermost ring is 1 point, a total of 10 rings. Rings with a score of 7-10 are made of black, and rings with a score of less than 7 are made of light cardboard. As the place where the diabol(bullet of the airpistol) hits moves away from the center, the score from the shot decreases. Shooting scoring; It is obtained by adding the points received for each shot by the Electronic Scoring System. Athletes should make 60 shots in 75 minutes. In this way, the total success score was calculated for each athlete. While 0 is the lowest score 600 is the highest score.
Shooting Performance | week 9
  Shooting performance will be calculated with electronic scoring system. (SIUS LS10 Laserscore, Swiss). Electronic Scoring System is an electronic target system for airguns. The target sign at which the shooting is made is 17x17 cm in size; The black dot with a diameter of 11.5 millimeters in the center is 10 points, and the outermost ring is 1 point, a total of 10 rings. Rings with a score of 7-10 are made of black, and rings with a score of less than 7 are made of light cardboard. As the place where the diabol(bullet of the airpistol) hits moves away from the center, the score from the shot decreases. Shooting scoring; It is obtained by adding the points received for each shot by the Electronic Scoring System. Athletes should make 60 shots in 75 minutes. In this way, the total success score was calculated for each athlete. While 0 is the lowest score 600 is the highest score.

SECONDARY OUTCOMES:
Shoulder abductor and adductor concentric muscle strength | baseline
  For shoulder abduction and adduction muscle strength, the athlete will be asked to perform 5 repetitions with maximal effort at an angular speed of 60°/sec.Shoulder abductor and adductor concentric muscle strengths will be measured with an isokinetic dynamometer. (Cybex Humac Norm Testing & Rehabilitation System, USA)
Shoulder abductor and adductor concentric muscle strength | week 9
  For shoulder abduction and adduction muscle strength, the athlete will be asked to perform 5 repetitions with maximal effort at an angular speed of 60°/sec.Shoulder abductor and adductor concentric muscle strengths will be measured with an isokinetic dynamometer. (Cybex Humac Norm Testing & Rehabilitation System, USA)
Shoulder abductor and adductor isometric muscle Strength | baseline
  For isometric muscle strength, contractions of 10 seconds will be required, with 5 repetitions in the direction of abduction and adduction at a 90° shoulder abduction angle.Shoulder abductor and adductor isometric muscle strengths will be measured with an isokinetic dynamometer. (Cybex Humac Norm Testing & Rehabilitation System, USA)
Shoulder abductor and adductor isometric muscle Strength | week 9
  For isometric muscle strength, contractions of 10 seconds will be required, with 5 repetitions in the direction of abduction and adduction at a 90° shoulder abduction angle.Shoulder abductor and adductor isometric muscle strengths will be measured with an isokinetic dynamometer. (Cybex Humac Norm Testing & Rehabilitation System, USA)
Upper extremity strength and endurance | baseline
  It will be evaluated by closed kinetic chain upper extremity test. Change in the number of touching hand number.
Upper extremity strength and endurance | week 9
  It will be evaluated by closed kinetic chain upper extremity test. Change in the number of touching hand number.
Scapular muscle endurance | baseline
  It will be evaluated by scapular muscle endurance test- Change in the time holding test position. A 10 Newton dynamometer will be used for the scapular muscle endurance test (Edulab, dynamometer, Turkey).
Scapular muscle endurance | week 9
  It will be evaluated by scapular muscle endurance test- Change in the time holding test position. A 10 Newton dynamometer will be used for the scapular muscle endurance test (Edulab, dynamometer, Turkey).
Core endurance-Unilateral Wall Sit Hold | baseline
  Change in the time holding.
Core endurance-Unilateral Wall Sit Hold | week 9
  Change in the time holding.
Core endurance-Trunk Flexion Hold | baseline
  Change in the time holding trunk flexion position. A standard goniometer will be used to establish proper positioning of the participant for each core test. Hold time duration wilk be recorded by the stopwatch feature on the raters' iPhones (Apple, Inc., Cupertino, CA).
Core endurance-Trunk Flexion Hold | week 9
  Change in the time holding trunk flexion position. A standard goniometer will be used to establish proper positioning of the participant for each core test. Hold time duration wilk be recorded by the stopwatch feature on the raters' iPhones (Apple, Inc., Cupertino, CA).
Core endurance-Horizontal Trunk Flexion Hold | baseline
  Change in the time holding horizontal trunk flexion position.A standard goniometer will be used to establish proper positioning of the participant for each core test. Hold time duration wilk be recorded by the stopwatch feature on the raters' iPhones (Apple, Inc., Cupertino, CA).
Core endurance-Horizontal Trunk Flexion Hold | week 9
  Change in the time holding horizontal trunk flexion position.A standard goniometer will be used to establish proper positioning of the participant for each core test. Hold time duration wilk be recorded by the stopwatch feature on the raters' iPhones (Apple, Inc., Cupertino, CA).

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No